CLINICAL TRIAL: NCT06157008
Title: Brain Network Analysis of Anesthesia Characteristics in Patients With Prolonged Disorders of Consciousness Based on Polysomnography
Brief Title: Brain Network Analysis of Anesthesia Characteristics in Patients With pDoC Based on PSG
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Other Study IDs: evchen99525
Record Dates: First submitted 2023-01-12; First posted 2023-12-05 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Anesthetics, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers
- patients with prolonged disorders of consciousness
  Interventions: Drug: General Anesthetics

INTERVENTIONS:
Drug: General Anesthetics — General anesthetics used in spinal cord electrical stimulator insertion surgery
  Groups: patients with prolonged disorders of consciousness

SUMMARY:
The goal of this prospective, exploratory and observational study is to learn about in healthy volunteers and patients with prolonged disorders of consciousness(pDoC). The main questions it aims to answer are:

1. Observe the similarities and differences of polysomnography between pDoC patients and healthy volunteers, and analyze the characteristic brain network changes based on polysomnography
2. To observe the similarities and differences of polysomnography in pDoC patients before and after Insertion of spinal cord electric stimulator under general anesthesia,and analyze the changes of anesthesia characteristic brain network in patients with consciousness disorders based on polysomnography.
3. To observe the similarities and differences of polysomnography in pDoC patients before and after spinal cord stimulation,and analyze the characteristic changes of brain network after spinal cord stimulation.

We will record the 8h polysomnography of healthy volunteers,record the polysomnography of DOC patients before and 24 hours after operation;and record the 24h polysomnography of patients with spinal cord electric stimulator.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria of health volunteer group:

  1. Aged 18-65, native Chinese
  2. No history of sleep apnea
  3. No history of insomnia
  4. Volunteer to participate in this study and obtain informed consent.
* Inclusion criteria of pDoC group:

  1. Aged 18-65, native Chinese
  2. pDoC after acquired brain injury
  3. The spinal electric stimulator was implanted under general anesthesia
  4. Obtain informed consent.
* Exclusion Criteria:

  1. Healthy volunteers took hypnotic drugs 72 hours before the study
  2. Continuous sedation treatment was carried out within 72 hours before the study
  3. The integrity of brain structures such as open head injury and brain parenchyma resection
  4. Intracranial compliance decreased due to hydrocephalus
  5. Airway stenosis and severe ventilation or ventilation dysfunction caused by various reasons
  6. Known or suspected to have serious heart, lung and kidney dysfunction
  7. Allergic history of sedative drugs
  8. Combined with other mental or nervous system diseases
  9. Other reasons are not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The people with prolonged disorders of consciousness who will be implanted with spinal cord electric stimulator under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of sleep in pDoC patients | January 1, 2023 to January 1, 2024
  Characteristics of sleep in pDoC patients compared with healthy volunteers
Sleep EEG and characteristic brain network in pDoC patients before and after anesthesia | January 1, 2023 to January 1, 2024
Sleep electroencephalogram and characteristic brain network of pDoC patients before and after starting the spinal cord electric stimulator | January 1, 2023 to January 1, 2024
Consciousness recovery of patients with pDoC 30 days, 90 days and 180 days after operation | January 1, 2023 to January 1, 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China